CLINICAL TRIAL: NCT01497197
Title: A Phase IIIb, Interventional, Multicentre, Multinational, Randomised, Open-label Trial to Compare the Efficacy and Safety of Ovarian Stimulation With GONAL-f® and Luveris® Starting on Day 1 vs. Day 6 in Women Between 36 and 42 Years of Age Undergoing Assisted Reproductive Technique (ART)
Brief Title: A Trial to Compare the Efficacy and Safety of Ovarian Stimulation With GONAL-f® and Luveris® Starting on Day 1 Versus Day 6 in Women Undergoing Assisted Reproductive Technique
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated as per sponsor's decision
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Middle East FZ LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EMR200061-506
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-10

CONDITIONS: Infertility; Fertility; Follicle Stimulating Hormone Deficiency
Keywords: Reproduction Techniques; Reproductive Medicine; Assisted Reproductive Technics; Pregnancy Rate; Ovulation Induction; Ovarian Stimulation; Oocytes; Implantation
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Luteinizing Hormone, beta Subunit; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gonal-f®+Luveris® (Experimental): GONAL f® 300 international units [IU] per day as subcutaneous injection using liquid pen from stimulation Day 1-5 followed by Luveris® 150 IU per day lyophilized powder for subcutaneous injection from stimulation Day 1 until required recombinant human chorionic gonadotropin (r-hCG) level is met. The dose will be adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the center's standard practice.
  Interventions: Drug: GONAL-f®; Drug: Luveris®; Biological: Recombinant human chorionic gonadotropin (r-hCG)
- Gonal-f® Followed by Luveris® (Experimental): GONAL-f® 300 IU per day as subcutaneous injection using liquid pen from stimulation Day 1-5 followed by Luveris® 150 IU per day lyophilized powder for subcutaneous injection from stimulation Day 6 until required r-hCG level is met. The dose will be adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the center's standard practice.
  Interventions: Drug: GONAL-f®; Drug: Luveris®; Biological: Recombinant human chorionic gonadotropin (r-hCG)

INTERVENTIONS:
Drug: GONAL-f® — GONAL f® 300 international units [IU] per day as subcutaneous injection using liquid pen.
Drug: Luveris® — Luveris® 150 IU per day lyophilized powder for subcutaneous injection.
Biological: Recombinant human chorionic gonadotropin (r-hCG) — A single injection of r-hCG (Ovidrel®/Ovitrelle®) 250 mcg to induce final oocyte maturation.

SUMMARY:
This is a phase IIIb, interventional, multicenter, multinational, randomised, open-label, comparative trial which primary objective is to generate data on the ovarian stimulation profile obtained when Luveris® is started either on Day 1 or Day 6 in women in advanced reproductive age (36-42) undergoing Assisted Reproductive Technique (ART).

DETAILED DESCRIPTION:
The subjects who complete the screening assessments and fulfil all the eligibility criteria will start down-regulation treatment on day 21-22 of the cycle.

Down-regulation treatment must start within 2 months following the screening visit. The routine long luteal phase protocol for Gonadotrophin-releasing hormone (GnRH) agonist treatment will be followed.

Once down-regulation has been confirmed, a pregnancy test will be performed within 1 week prior to start of Recombinant human follicle stimulating hormone (r-hFSH) treatment to rule out any pre-existing pregnancy. If the result is negative, the subject will be randomly assigned to one of the two treatment arms of the trial:

* GONAL-f® (Liquid Pen; 300 IU of per day) stimulation day 1-5 then followed by Luveris® (vial/powder, 150 IU per day) from stimulation Day 1 and until required r-hCG level is met. The dose can be adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the center's standard practice.
* GONAL-f® (Liquid Pen; 300 IU per day) stimulation Day 1-5 then add Luveris® (vial/powder, 150 IU per day) from stimulation Day 6 and until required recombinant Human chorionic gonadotrophin (r-hCG) level is met. The dose can be adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the center's standard practice.

Randomization across the two treatment arms will be kept balanced in a 1:1 ratio. Subjects will be provided with a subject diary (including r-hCG and Crinone® administration and safety information) to record daily dosing information for GONAL-f® and Luveris®.

Follicular development will be monitored according to the center's standard practice by US and/or Oestradiol (E2) levels, until the protocol r-hCG requirement is met (i.e., at least 1 follicle greater or equal to 18 mm and 2 follicles greater or equal to 16 millimeter [mm]). After this, a single injection of 250 microgram (mcg) of r-hCG (Ovidrel®/Ovitrelle®), will be administered in order to induce final oocyte maturation.

At a time of 34-38 hours after r-hCG administration, oocytes will be recovered vaginally under US monitoring. Oocytes will then be fertilized in vitro and embryos replaced 2-3 days after oocyte recovery. Ovum pick up (OPU), in vitro fertilization (IVF), Embryo Transfer (ET) and luteal support will be performed as per center's standard practice. In addition, Crinone® 8% (progesterone gel) will be administered once daily.

A post-treatment safety visit will be performed for all subjects who received r-hCG (pregnant and non-pregnant) on post r-hCG Day 15-20. For subjects who have withdrawn from treatment (i.e. after starting Luveris® or GONAL f® but before r-hCG is given) this visit will take place 20-30 days after their first Luveris® or GONAL-f® treatment injection (excluding pregnancy testing).

ELIGIBILITY:
Inclusion Criteria:

* Should be a female subject justifying an In Vitro Fertilization/Embryo transfer (IVF)/ET treatment
* Should be between 36th and 42nd birthday (both included) at the time of the randomization visit
* Have early follicular phase (day 2-4) serum level of basal FSH <= 12 IU/L measured in the center's local laboratory during the screening period (i.e. within 2 months prior to down regulation start)
* Have a regular spontaneous ovulatory menstrual cycle between 21 and 35 days in length
* Presence of both ovaries
* Normal uterine cavity, which in the investigator's opinion is compatible with Pregnancy
* Have a negative cervical Papanicolaou (PAP or smear) test within the last 6 months prior to randomization
* Have at least one wash-out cycle (defined as >=30 days since the last dose of clomiphene citrate or gonadotrophin treatment) since the last ART cycle and/or clomiphene citrate or gonadotrophin treatment prior to starting GnRH agonist therapy
* Be willing and able to comply with the protocol for the duration of the trial
* Have given written informed consent, prior to any trial-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to her future medical care
* Have a male partner with semen analysis within the past 6 months prior to randomization considered adequate to proceed with regular insemination or intra-cytoplasmic sperm injection (ICSI) according to the center's standard practice

Exclusion Criteria:

* Had 2 (or more) previous ART cycles with a poor response to gonadotrophin stimulation defined as 6 (or less) mature follicles and/or 4 (or less) oocytes collected in any previous IVF cycle or previous cycles with a hyper response defined as 25 (or more) oocytes retrieved
* Any medical condition, which in the judgment of the investigator may interfere with the absorption, distribution, metabolism or excretion of the drug. In case of doubt, the subject in question should be discussed with Merck Serono's Medical responsible
* Had previous severe ovarian hyperstimulation syndrome (OHSS)
* Polycystic ovary syndrome (PCOS; Rotterdam criteria) to reduce the risk of the occurrence of OHSS
* Presence of endometriosis requiring treatment
* Uterine myoma requiring treatment
* Any contraindication to being pregnant and/or carrying a pregnancy to term
* Extra-uterine pregnancy within the last 3 months prior to screening
* History of 3 or more miscarriages (early or late miscarriages) due to any cause
* Tumours of the hypothalamus and pituitary gland
* Ovarian enlargement or cyst of unknown etiology
* Ovarian, uterine or mammary cancer
* A clinically significant systemic disease
* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or C virus in the trial subject or her male partner
* Abnormal gynecological bleeding of undetermined origin
* Known allergy or hypersensitivity to human gonadotrophin preparations
* Any active substance abuse or history of drug, medication or alcohol abuse in the past 5 years prior to the screening visit
* Entered previously into this trial or simultaneous participation in another clinical trial
* Pregnancy and lactation period
* Participation in another clinical trial within the past 30 days

Ages: 36 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Serono Middle East FZ LLC
Locations (1):
- Merck Serono Research Site, Dubai, United Arab Emirates

RESULTS

PARTICIPANT FLOW:
Groups:
- Gonal-f®+Luveris: GONAL f® (Liquid Pen; 300 international units [IU] of per day) stimulation Day 1-5 then followed by Luveris® (vial/powder, 150 IU per day) from stimulation Day 1 until required r-hCG level was met. The dose was adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the centre's standard practice.
- Gonal-f® Followed by Luveris: GONAL-f® (Liquid Pen; 300 IU per day) stimulation Day 1-5 then added Luveris® (vial/powder, 150 IU per day) from stimulation day 6 until required r-hCG level was met. The dose was adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the centre's standard practice.
Period: Overall Study
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Started | 89 | 85
Completed | 72 | 70
Not Completed | 17 | 15
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Excessive/lack of response to treatment | 1 | 0
Not completed — Risk of OHSS | 1 | 0
Not completed — No oocytes retrieved | 3 | 2
Not completed — No fertilisation | 6 | 5
Not completed — Intention to freeze all embryos | 0 | 1
Not completed — All embryos discarded | 0 | 3
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all the subjects randomized in the study.
Groups:
- Gonal-f®+Luveris: GONAL f® 300 international units [IU] per day as subcutaneous injection using liquid pen from stimulation Day 1-5 followed by Luveris® 150 IU per day lyophilized powder for subcutaneous injection from stimulation Day 1 until required recombinant human chorionic gonadotropin (r-hCG) level was met. The dose was adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the center's standard practice.
- Gonal-f® Followed by Luveris: GONAL-f® 300 IU per day as subcutaneous injection using liquid pen from stimulation Day 1-5 followed by Luveris® 150 IU per day lyophilized powder for subcutaneous injection from stimulation Day 6 until required r-hCG level was met. The dose was adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the center's standard practice.
- Total: Total of all reporting groups
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris | Total
Number analyzed (Participants) | 89 | 85 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (1.6) | 38 (1.7) | 37.9 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 85 | 174
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Oocytes Retrieved Per Subject Following Ovarian Stimulation
Description: Ovarian stimulation was performed using in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI). The total number of oocytes collected per subject following stimulation was reported.
Time Frame: 34-38 hours post r-hCG administration
Population: Modified intention-to-treat (MITT) included all the subjects randomized into the trial who received at least 1 dose of Gonal-f® or Luveris®, and who completed the primary efficacy assessment (total number of oocytes retrieved per subject following recombinant human follicle stimulating hormone (r-hFSH) stimulation and r-hCG injection).
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 86 | 82
oocytes | 8.6 (6.54) | 8.7 (5.77)

2. Secondary Outcome: Total Dose and Mean Daily Dose of Follicle Stimulating Hormone (FSH)
Description: Mean daily dose of FSH was to be determined by dividing the total daily dose by the number of stimulation days.
Time Frame: Screening
Population: Data was not analysed as per planned analysis due to frequent protocol violations/deviations, there was no subject eligible to be analyzed per protocol.
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Total Number of Stimulation Treatment Days
Description: The total number of stimulation treatment days for each subject was determined based on the treatment administration information collected in the case report form.
Time Frame: 6 days post stimulation (Number of stimulation days+6 days)
Population: MITT included all the subjects randomized into the trial who received at least 1 dose of Gonal-f® or Luveris®, and who completed the primary efficacy assessment (total number of oocytes retrieved per subject following r-hFSH stimulation and r-hCG injection).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 86 | 82
days | 11.1 (2.42) | 11.3 (2.24)

4. Secondary Outcome: Implantation Rate
Description: The implantation rate was determined as number of fetal sacs divided by the number of embryos transferred post r-hCG administration.
Time Frame: 35-42 days post r-hCG administration
Population: MITT included all subjects randomized in the trial who received at least 1 dose of Gonal-f® or Luveris®, and who completed primary efficacy assessment(total number of oocytes retrieved/subject following r-hFSH stimulation and r-hCG injection). 'N' signifies all subjects who showed positive pregnancy test and evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: fetal sacs/embryo transferred
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 19 | 21
fetal sacs/embryo transferred | 0.5 (0.51) | 0.4 (0.51)

5. Secondary Outcome: Number of Fetal Sacs With Activity
Description: Number of fetal sacs with activity was evaluated by ultrasound scan (US) on Days 35-42 post r-hCG to confirm clinical pregnancy.
Time Frame: 35-42 days post r-hCG administration
Population: MITT included all subjects randomized in the trial who received at least 1 dose of Gonal-f® or Luveris®, and who completed primary efficacy assessment(total number of oocytes retrieved/subject following r-hFSH stimulation and r-hCG injection). 'N' signifies all participants who showed positive pregnancy test and evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Fetal sacs
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 19 | 21
Fetal sacs | 0.8 (0.42) | 1.1 (0.54)

6. Secondary Outcome: Number of Fetal Sacs With Detectable Heart Beats
Description: Number of fetal sacs with detectable heart beats was evaluated by US on Days 35-42 post r-hCG to confirm clinical pregnancy
Time Frame: 35-42 days post r-hCG administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Fetal sacs
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 19 | 21
Fetal sacs | 0.6 (0.50) | 1.0 (0.45)

7. Secondary Outcome: Total Pregnancy Rate and Clinical Pregnancy Rate
Description: The subject was considered to have a positive pregnancy result if beta-hCG >10 international units per liter (IU/L) and the subject had not menstruated between post-r-hCG Days 15-20. Clinical pregnancy was defined as the existence of at least an US confirmed gestational sac in the uterus with fetal heart activity post-r-hCG Days 35-42.
Time Frame: 35-42 days post r-hCG administration
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 86 | 82
percentage of subjects
  Total pregnancy | 20 | 27
  Clinical pregnancy | 17 | 23

8. Secondary Outcome: Cycle Cancellation Rate Prior to r-hCG
Description: If the subject was not administered with r-hCG and withdrew prematurely from the trial, it was considered as cycle cancellation.
Time Frame: Up to 85 days
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 86 | 82
percentage of subjects | 0 | 0

9. Secondary Outcome: Number of Subjects With Biochemical Pregnancies
Description: Biochemical pregnancy was defined as the pregnancy diagnosed only by the detection of hCG in serum or urine and that does not develop into a clinical pregnancy. Subjects with beta-hCG concentration greater than 10 IU/L were considered as biochemical pregnant.
Time Frame: 35 to 42 days post r-hCG administration
Population: as for outcome 3
Measure: Number; unit: subjects
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 86 | 82
subjects | 2 | 1

10. Secondary Outcome: Number of Subjects With Multiple Pregnancies
Description: Multiple pregnancy was defined as the existence of more than one ultrasound confirmed gestational sac in the uterus with fetal heart activity at post-r-hCG Days 35-42.
Time Frame: 35 to 42 days post r-hCG administration
Population: MITT included all subjects randomized into trial who received at least 1 dose of Gonal-f® or Luveris®, and completed the primary efficacy assessment (total number of oocytes retrieved per subject following r-hFSH stimulation and r-hCG injection). 'N'=signifies all subjects who showed positive pregnancy test and evaluable for this outcome measure.
Measure: Number; unit: subjects
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 19 | 21
subjects | 0 | 4

11. Secondary Outcome: Number of Subjects With Any Adverse Events (AEs), Serious AEs, AEs Leading to Death, and AEs Leading to Discontinuation
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A serious AE is an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Baseline up to 15-20 days post r-hCG administration
Population: Safety population included all randomized subjects who received at least one dose of the trial treatment.
Measure: Number; unit: subjects
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Number analyzed (Participants) | 89 | 85
subjects
  AEs | 27 | 28
  Serious AEs | 4 | 5
  AEs Leading to Death | 0 | 0
  AEs Leading to Discontinuation | 1 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to 15-20 days post r-hCG administration
Arm/Group | Gonal-f®+Luveris | Gonal-f® Followed by Luveris
Serious Adverse Events (participants affected / at risk) | 4/89 | 5/85
Other Adverse Events (participants affected / at risk) | 24/89 | 27/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gonal-f®+Luveris (N=89) | Gonal-f® Followed by Luveris (N=85)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 4
Ovarian cyst (Reproductive system and breast disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gonal-f®+Luveris (N=89) | Gonal-f® Followed by Luveris (N=85)
Overdose (Injury, poisoning and procedural complications) | 13 | 14
Oestradiol increased (Investigations) | 8 | 8
Progesterone increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 5
Breast pain (Reproductive system and breast disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated as per sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less